CLINICAL TRIAL: NCT06745674
Title: Effectiveness of Internet-based Acceptance and Commitment Therapy for Cancer Patients: A Pilot Randomized Controlled Trial Using Mixed Methods
Brief Title: Online Intervention for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Centrl China Normal University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-202311017b
Record Dates: First submitted 2024-12-08; First posted 2024-12-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist control group (No Intervention)
- ACT group (Experimental)
  Interventions: Behavioral: a mobile app-delivered Acceptance Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: a mobile app-delivered Acceptance Commitment Therapy (ACT) — The study utilized a specially tailored internet-based self-help ACT program for cancer patients. It consisted of an introductory module and six core intervention modules: (1) Refusing Avoidance; (2) Accepting Distress; (3) Living in the Present Moment; (4) Observing Yourself Psychologically; (5) Exploring Meaningful Values; and (6) Committing to Action. Each module, designed to take 30-60 minutes, was delivered over a two-week period.
  Arms: ACT group

SUMMARY:
This study will focus on supporting cancer patients who often experience emotional challenges like anxiety and depression. It will test a two-week online program called Acceptance and Commitment Therapy (ACT), designed to help people manage difficult emotions and focus on what matters most in their lives.

The program will include short, easy-to-follow sessions covering helpful strategies like accepting distress and staying present in the moment. Participants will be randomly assigned to either join the ACT program or wait for the program while continuing their usual care. The study aims to determine whether the ACT program can reduce psychological distress, anxiety, and depression in cancer patients. The study will use a mixed-methods approach, combining both quantitative data (such as changes in distress, anxiety, and depression) and qualitative insights from participant interviews. This will help us gain a deeper understanding of how the ACT program may support the psychological distress of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above;
* diagnosed cancer with a clear disease course
* fluent in Chinese with the ability to read and understand questionnaires independently;
* ability to operate a smartphone independently;
* not participating in or intervening in other clinical studies.

Exclusion Criteria:

* younger than 18 years of age
* unable to use a smartphone
* have significant cognitive impairment or a serious systemic disease or psychiatric disorder
* concurrently participating in other clinical studies or undergoing other psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility outcomes | Post-intervention (immediately after the 2-week intervention)
  Feasibility is evaluated using retention rate and intervention completion rate. Retention rate reflects the percentage of participants who successfully completed all study-related measurements throughout the trial.
Psychological Distress | Baseline, one week post-baseline, and post-intervention (immediately after the 2-week intervention)
  Psychological distress is assessed using the Distress Thermometer (DT) (Holland et al., 2013). Scores range from 0 (no distress) to 10 (extreme distress), with higher scores reflecting greater levels of psychological distress.
Anxiety and Depression | Baseline, one week post-baseline, and post-intervention (immediately after the 2-week intervention)
  Anxiety and depression are measured using the Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983), a 14-item questionnaire comprising separate subscales for anxiety and depression. Each item is scored on a 4-point Likert scale, and higher scores reflect greater severity of anxiety and depression symptoms.
Acceptability | Post-intervention (immediately after the 2-week intervention)
  Acceptability is evaluated using the Client Satisfaction Questionnaire (CSQ-8) (Larsen et al., 1979). This 8-item measure uses a 4-point Likert scale (1 = low satisfaction to 4 = high satisfaction), with higher scores indicating greater satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes